CLINICAL TRIAL: NCT06466265
Title: An Open-label, Dose-finding, Phase I Study to Assess the Safety, Tolerability, and Pharmacokinetic Profile of DNP002 in Patients With Advanced Solid Tumors
Brief Title: Study of DNP002 in Patients With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kumho HT Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCC2021-0034
Record Dates: First submitted 2024-06-12; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant Group/Arm (Experimental): Experimental: Patients with advanced solid tumors
  Dose escalation with patients having solid tumors. Patients receive escalating doses of DNP002 intravenously for 1 hour on Day 1 of each 14-day cycle (Q2W) or each 21-day cycle (Q3W).
  This course will be repeated in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: DNP002

INTERVENTIONS:
Drug: DNP002 — Anti-CEACAM6 monoclonal antibody
  Other Names: H2319

SUMMARY:
This is an open-label, Phase 1, first-in-human, dose-escalation study designed to assess the safety, tolerability, pharmacokinetics, and preliminary efficacy of the anti-Carcinoembryonic-antigen-related-cell-adhesion-molecule-6 (CEACAM6) antibody DNP002 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
The primary objectives of this study are to evaluate the safety and tolerability of DNP002 in patients with advanced solid tumors, and to determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D). The secondary objectives are to evaluate the pharmacokinetic properties and preliminary anti-tumor effects in patients with solid tumors. The exploratory objectives are to analyze the expression and relationship with efficacy of various tumor and blood biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 19 years or older as of the date of written informed consent.
2. Patients with histologically or cytologically confirmed unresectable locally advanced and/or metastatic solid tumors who have been refractory to or had disease progression after standard treatment and have no other available standard treatment options.
3. Patients with at least one measurable or evaluable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
4. Patients with an expected survival of greater than or equal to 12 weeks.
5. Patients with Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
6. Patients confirmed to have adequate hematologic, renal, and hepatic function.
7. Patients who have recovered to National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade 1 or baseline status from reversible side effects of prior anticancer therapies (excluding alopecia [regardless of grade] or grade 2 peripheral neuropathy or any laboratory test, blood pressure, and ECG results that meet the inclusion/exclusion criteria).
8. For women of childbearing potential, negative pregnancy test (urine-hCG and/or serum hCG) at the time of clinical trial participation.
9. For women of childbearing potential and men, no plans for pregnancy from screening to 24 weeks after treatment cessation and willingness to use appropriate contraception methods.
10. Voluntary written informed consent for clinical trial participation.

Exclusion Criteria:

1. At the screening visit, you have any of the following comorbidities:

1. Hematologic malignancies, including lymphoma.
2. Interstitial lung disease or pulmonary fibrosis.
3. Bowel obstruction or bowel perforation.
4. Clinically significant pleural effusion, ascites, or pleural effusion.
5. Severe infections or other uncontrolled active infectious diseases requiring treatment with antibiotics, antiviral drugs, etc. that may affect safety and efficacy evaluation during the clinical trial period, as determined by the investigator.
6. Uncontrolled hypertension (systolic blood pressure (SBP) /diastolic blood pressure (DBP) ≥ 160/100 mmHg).
7. QTc interval exceeding 480 msec (same criteria for both sexes) using Fridericia's QT correction formula.
8. Active hepatitis B or C (hepatitis C virus antibody (HCV Ab) positive but HCV ribonucleic acid (RNA) negative may be considered as previous infection and eligible for clinical trial).
9. Clinically significant symptoms or uncontrolled central nervous system (CNS) metastases or carcinomatous meningitis (clinical trial eligibility is possible if no progression has been confirmed clinically and on computed tomography (CT)/magnetic resonance imaging (MRI) for at least 4 weeks prior to the administration of investigational drugs after treatment for CNS or brain metastases and no treatment with steroids or other medications is required at least 2 weeks before administration of investigational drugs).

2. At the screening visit, individuals with the following medical history (including surgical/intervention history):

1. Major surgery or clinically significant traumatic injury within 4 weeks prior to screening
2. Significant cardiovascular disease such as unstable angina, myocardial infarction, congestive heart failure, stroke, or unstable arrhythmia within 24 weeks prior to screening
3. Immunosuppressive disease (e.g., acquired immune deficiency syndrome (AIDS), human immunodeficiency virus (HIV), etc.) or autoimmune disease
4. Psychiatric disorder that, in the opinion of the investigator, significantly affects the clinical trial

3. Subjects who have received the following drug therapies (pharmacological/non-pharmacological):

1. History of immunosuppressive medication within 2 weeks prior to baseline (Day 1 administration date) (Note: Topical, ophthalmic, intra-articular, intranasal, inhaled corticosteroids, and systemic corticosteroids with prednisolone equivalent to 10 mg/day or less are considered exceptions)
2. Other anticancer therapy (excluding investigational medicinal products and immune checkpoint inhibitors) within 3 weeks prior to baseline (Day 1 administration date) (Note: Point radiation for the purpose of relieving symptoms such as bone pain, bronchial obstruction, and skin lesions is allowed, but participation is not allowed if the subject has a history of nitrosoureas or mitomycin-C within 6 weeks prior to baseline)

   *Radiation (chemo)therapy, chemotherapy, targeted agents (small molecule drugs, monoclonal antibodies), hormonal therapy, etc.
3. History of immune checkpoint inhibitor administration within 4 weeks prior to baseline (Day 1 administration date) (e.g., anti-programmed cell death protein 1 (PD-1), anti-programmed death-ligand 1 (PD-L1), anti-PD-L2, anti-cluster of differentiation (CD) 137, anti-cytotoxic T-lymphocyte associated protein 4 (CTLA-4), etc.)
4. History of anti-carcinoembryonic antigen-related cell adhesion molecule (CEACAM) 6 medication within 4 weeks prior to baseline (Day 1 administration date)

4. Subjects with severe hypersensitivity or other immune-related adverse events to monoclonal antibody preparations or the active substance or excipients of DNP002

5. Subjects who participated in other clinical trials and received investigational products (or medical devices) within 4 weeks prior to baseline

6. Other subjects who are deemed ineligible for this clinical trial by the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | Up to 2 or 3 weeks
  DLT is assessed according to NCI-CTCAE v5.0. The assessment is conducted only in the 2-week interval for subjects receiving the first dose (2-week interval subject) or the 3-week interval for subjects receiving the first dose (3-week interval subject).
Incidence and severity of treatment emergent adverse events | Up to 2 years
  Describe the character and incidence of toxicity based on CTCAE v5.0 that occur receiving DNP002.
Characterize the area under the concentration-time curve (AUC) of the pharmacokinetics (PK) of DNP002 | Day 1 (pre-dose), 1 hour (post-dose), 2, 4, 8 10, 12 hours, Day 2, Day 3, Day 8 after 1st or 5th doses of the investigational drug.
  Samples for pharmacokinetic evaluation will be collected immediately prior to each of the 5 doses, and at predetermined time intervals after the 1st and 5th doses.
Characterize peak plasma concentration (Cmax) of the pharmacokinetics (PK) of DNP002 | Day 1 (pre-dose), 1 hour (post-dose), 2, 4, 8 10, 12 hours, Day 2, Day 3, Day 8 after 1st or 5th doses of the investigational drug.
  Samples for pharmacokinetic evaluation will be collected immediately prior to each of the 5 doses, and at predetermined time intervals after the 1st and 5th doses.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years
  Percentage of patients whose best response to DNP002 is either a Complete response or Partial response, both defined according to RECIST or iRECIST criteria respectively.
Leukocyte immune phenotyping | Day 1 (pre-dose), before the first, third, and fifth doses of the investigational drug, as well as 24 hours after the first and fifth doses.
  Whole blood flow cytometry analysis for characterization of blood leukocyte/lymphocyte including MDSC with regards to subpopulation and activation before and under treatment in all patients.
Serum biomarkers | Day 1 (pre-dose), before the first, third, and fifth doses of the investigational drug, as well as 4 hours after the first and fifth doses.
  Total concentration of Arginase-1, soluble CEACAM6, CEA, Interferon-gamma and Interleukin-6 in serum derived from whole blood taken before and under treatment in all patients.
Concentration of anti-drug antibodies | Prior to administration at each dose (The investigational drug should be continued with dosing every two weeks as long as there is no disease progression or unacceptable toxicity.)
  Concentration in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Moonki Choi, M.D., Ph.D., Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea